CLINICAL TRIAL: NCT01849705
Title: Mutations in the Melanocortin 4 Receptor and Obesity-associated Diseases
Brief Title: Melanocortin 4 Receptor Mutations and Obesity-associated Diseases
Acronym: Mc4Obes
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, AAstrup, MD, Professor, University of Copenhagen
Other Study IDs: B-298; H-2-1012-108 (Registry Identifier: The Danish National Committee on Biomedical Research Ethics)
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: Obesity; MC4R; Blood pressure; Blood glucose
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Mutations in the melanocortin 4 receptor (MC4R) are the most common form of monogenic obesity, and can explain 2-6% of severe obesity.

Studies have shown that mutations in MC4R are associated with increased fat mass, height-for-age, appetite and insulin resistance among children. In adults, mutations in MC4R are less penetrant for these phenotypes but it has been observed that individuals with MC4R mutations have a smaller than expected blood pressure for their degree of obesity.

The purpose of this study is to explore the association between functional MC4R mutations and obesity, insulin resistance and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Men and women
* BMI > 30 kg/m^2

Exclusion Criteria:

* Uncontrolled type 2 diabetes
* Bariatric surgery
* Use of anti-obesity medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18-70 years
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure | Baseline
  Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Obesity | Baseline
  Obesity measured as BMI
Blood glucose | Baseline
  Blood glucose measured at baseline
MC4R mutations | Baseline
  MC4R mutations detected by sequencing of the coding region of the MC4R gene

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, MD, Dr. Med, Study Director — Department of Human Nutrition, University of Copenhagen; Lesli H Larsen, PhD, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Frederiksberg, Frederiksberg C, Denmark